CLINICAL TRIAL: NCT06789055
Title: Efficacy of a Cold Spray in Reducing Pain During Capillary Glucose Testing: a Randomized Controlled Trial
Brief Title: Cold Spray's Role in Reducing Pain During Capillary Glucose Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Faruk Danış, MD, Principal Investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BAIBU-TF-FD-01
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Visual Analog Pain Scale
Keywords: Cold Spray; Capillary Glucose Testing; Pain Management; Patient Comfort
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized crossover trial. Patients requiring at least two capillary blood glucose measurements were included in the study. Participants were randomized into two groups. In the first group, placebo was applied during the first measurement, and cold spray was used for the second measurement. Conversely, in the second group, cold spray was applied prior to the first glucose measurement, followed by placebo during the second measurement. This crossover design ensures that each patient serves as their own control, minimizing inter-individual variability and enhancing the reliability of the findings.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other): In the first group, placebo will be applied prior to the initial capillary blood glucose measurement, after which the measurement will be performed, and the patient's pain level will be assessed using the Visual Analog Scale (VAS). For the subsequent second measurement, cold spray will be applied before the procedure, followed by the glucose measurement, which will be conducted on the same finger of the opposite hand as used in the first measurement. The patient's pain level will again be evaluated using the VAS. This sequential approach allows for a direct comparison of pain scores between placebo and cold spray applications within the same patient.
  Interventions: Other: Cold Spray; Other: Placebo
- Group 2 (Other): In the second group, cold spray will be applied prior to the initial capillary blood glucose measurement, after which the measurement will be performed, and the patient's pain level will be assessed using the Visual Analog Scale (VAS). For the subsequent second measurement, placebo will be applied before the procedure, followed by the glucose measurement, which will be conducted on the same finger of the opposite hand as used in the first measurement.. This sequential approach allows for a direct comparison of pain scores between placebo and cold spray applications within the same patient.
  Interventions: Other: Cold Spray; Other: Placebo

INTERVENTIONS:
Other: Cold Spray — Before the capillary blood glucose measurement, cold spray will be applied to the measurement site from a distance of 30 cm for 10 seconds. Following this, the area will be cleansed with an antimicrobial swab for 10 seconds using a circular motion, starting from the center and moving outward. Subsequently, the fingertip will be punctured with a lancet to obtain a blood sample. The first drop of blood will be wiped away with cotton, and the glucose measurement will be performed using the subsequent drop utilizing the Standard GlucoNavii GDH device. The patient will then be asked to assess their pain during the procedure using the Visual Analog Scale (VAS) for pain evaluation.
Other: Placebo — Before the capillary blood glucose measurement, placebo will be applied to the measurement site from a distance of 30 cm for 10 seconds. Following this, the area will be cleansed with an antimicrobial swab for 10 seconds using a circular motion, starting from the center and moving outward. Subsequently, the fingertip will be punctured with a lancet to obtain a blood sample. The first drop of blood will be wiped away with cotton, and the glucose measurement will be performed using the subsequent drop utilizing the Standard GlucoNavii GDH device. The patient will then be asked to assess their pain during the procedure using the Visual Analog Scale (VAS) for pain evaluation.

SUMMARY:
The goal of this clinical trial is to learn if applying a cold spray can reduce pain during capillary blood glucose measurements in adults aged 18 years or older who need at least two blood glucose tests. The main questions it aims to answer are:

Does cold spray reduce pain levels, as measured by the Visual Analogue Scale (VAS) for pain? How do pain levels compare between cold spray and placebo spray? Researchers will use a crossover design to compare a cold spray application to a placebo spray to see if there is a meaningful difference in pain reduction.

Participants will:

Receive both cold spray and placebo spray in a specific sequence Have their pain levels measured using the Visual Analogue Scale (VAS) for pain during each measurement.

DETAILED DESCRIPTION:
Background/Aim: Capillary blood glucose measurement is a common procedure in emergency departments for the assessment and management of metabolic conditions. Despite its routine nature, the skin puncture required for this procedure causes varying degrees of discomfort or pain for patients. Non-pharmacological approaches to pain management, such as the application of cold spray, offer a simple and cost-effective solution to enhance patient comfort and satisfaction. This study aims to investigate the effectiveness of cold spray in reducing pain during capillary blood glucose measurements.

Methodology:

This study is designed as a randomized controlled crossover trial. Each patient serves as their own control to minimize variability and improve the reliability of results.

Adults aged 18 years or older, who require at least two capillary blood glucose measurements for any reason and provide informed consent to participate in the study, will be included.

Patients will be randomized into two groups (details about randomisation and groups are given in the relevant section). In the intervention process: cold spray will be applied to the site of measurement from 30 cm for 10 seconds, followed by cleansing with an antimicrobial swab using a circular motion for another 10 seconds. For the placebo, sterile water will be applied in the same manner.

For both group the fingertip will then be punctured with a lancet, and the first drop of blood will be wiped away before obtaining the sample from the subsequent drop. Pain levels during the procedure will be assessed using the Visual Analog Scale (VAS), a 100-mm line ranging from "no pain" (0) to "severe pain" (100).

The primary outcome is the pain level recorded using the VAS after each capillary blood glucose measurement.

Significance: This study aims to provide evidence on the efficacy of cold spray as a non-pharmacological method to reduce pain during routine capillary blood glucose measurements. The findings may lead to improved patient comfort and satisfaction in emergency department settings, with potential implications for other routine procedures involving skin puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients requiring at least two capillary blood glucose measurements for any reason
* Patients who agree to participate in the study

Exclusion Criteria:

* Allergy to the components of the spray
* Conditions that may affect capillary blood glucose measurement or pain perception, such as peripheral neuropathy or peripheral arterial disease
* Blood glucose levels outside the measurable range of the capillary device (extremely low or high levels)
* Cognitive disorders that prevent the evaluation of the Visual Analog Scale (VAS), such as dementia, Alzheimer's disease, or cerebrovascular diseases
* Severe conditions in other parts of the body that may interfere with pain evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Immediately after blood glucose measurement, assessed within the first 5 minutes after the procedure.
  The primary outcome of this study is the Visual Analog Scale (VAS) score for pain. The VAS is a widely used assessment tool to evaluate variables across a continuum, such as acute pain severity. For the purpose of this study, patients will be presented with a 100-mm line, where one end is labeled "no pain" and the other end is labeled "severe pain." After each capillary blood glucose measurement, patients will be asked to mark their level of pain on the VAS line based on their experience during the procedure. The VAS score will be determined by measuring the distance in millimeters from the "no pain" end to the point marked by the patient. This standardized and validated method provides a quantitative measure of pain that is both simple and reliable for clinical use.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No